CLINICAL TRIAL: NCT07103590
Title: New Design Sagittal Split Plate Versus Two Miniplates in the Treatment of Mandibular Angle Fractures (Randomized Controlled Clinical Trial)
Brief Title: Sagittal Split Plate Versus Two Miniplates in the Treatment of Mandibular Angle Fractures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1026-1/2025
Record Dates: First submitted 2025-07-15; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental)
  Interventions: Procedure: single Sagittal Split plate
- Conventional Group (Active Comparator)
  Interventions: Procedure: two conventional miniplates

INTERVENTIONS:
Procedure: single Sagittal Split plate — patients will be treated using a single Sagittal Split plate at the neutral zone of mandible
  Arms: Test Group
Procedure: two conventional miniplates — patients will be treated using two conventional miniplates according to Champy's osteosynthesis lines.
  Arms: Conventional Group

SUMMARY:
Mandibular fractures are the second most common maxillofacial fracture after nasal bone fracture. As a result, a lot of research work has gone into improving treatment methods for these fractures including, reduction of immobilization period and enhancement of rigid fixation. One of these modalities is the use of Sagittal Split plate at the angle of the mandible.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from recent, uninfected angle mandibular fracture.
* Fracture that demands open reduction and internal fixation.

Exclusion Criteria:

* Medically compromised patients contradicting the operation.
* Existence of infection at the fracture line.
* Pathological fracture.
* An old fracture.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores | baseline, 24 hours, 1 week, and 6 weeks
  Will be assessed through a 10-point Visual Analogue Scale (VAS) (34). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe).
Change in Maximal Inter-Incisal Mouth | baseline, 24 hours, 1 week, and 6 weeks
  Using a millimeter ruler to measure maximal inter-incisal mouth opening

SECONDARY OUTCOMES:
postoperative infection | 24 hours, 1 week, and 6 weeks
  observation for any manifestations of wound healing disturbance
change in bone density | baseline and 12 weeks
  Immediate CT (T0) scan will be done and then another CT (T1) will be taken at 12th week to estimate the mean bone density at the fracture line in comparison with the immediate postoperative scan

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No